CLINICAL TRIAL: NCT04956029
Title: Comparing Visual Inspection, Performance Observation, and Aerobic Colony Counts for Evaluating Hospital Cleanliness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Chen Ying-Chun, infection control nurse, Taichung Veterans General Hospital
Other Study IDs: CW21156B
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Auditing Methods for Hospital Cleanliness
Keywords: visual inspection; performance observation; aerobic colony counts; hospital cleanliness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There are no any interventions. This is to observe and test hospital cleanliness. — There are no any interventions. This is to observe and test hospital cleanliness.

SUMMARY:
This study aims to compare correlation between outcome and performance observations and effectiveness by using aerobic colony counts as a comparator in order to find out which method would be better to be used to assess hospital cleanliness.

DETAILED DESCRIPTION:
Design and Setting We perform a prospective study which is conducted in a 17-bed adult medical intensive care unit with approximately 352 annually admissions at a tertiary hospital in Taiwan from July 2021 to December 2022. Cleaning performance observation will be performed according to the environmental checklist for monitoring terminal cleaning released by Centers for Disease Control and Prevention in 2014, to select sampling areas of high-touch surfaces in patient rooms, including bed controls, bed rails, cart pulls, light switches, machine controls, tray tables and call buttons.

Data collection The housekeepers start to do terminal cleaning after patients are transferred or discharged, the researcher also starts to observe directly the practices of cleaning at the same time and recorded "compliant" or "not compliant" whenever surfaces are cleaned and disinfected properly or on the contrary. The high-touch surfaces are disinfected with solution which contained Sodium dichloroisocyanurate (NaDCC). Right after the surfaces are cleaned, the researcher inspect the surfaces and record "clean" or "not clean" whenever surfaces are free of dust, debris, and stains immediately after terminal cleaning or on the contrary.

Ten minutes after surfaces are cleaned and disinfected, Hygiena Ultrasnap Surface ATP test will be applied to swab a standard 10*10 cm area on selected surfaces by samping templet. After completing sampling, swabs are replaced back in swab tube and all liquid in bulbs was expelled to activate the reaction. Once activated, samples were read right after shaking swab tube for 5-10 seconds. The ATP readings less than 10 RLU (relative light unit, RLU) are interpreted as "pass".

The designated cleaner and the researcher will be assigned to clean high-touch room surfaces and to be in charge of evaluating and sampling, respectively.

Statistical analysis Descriptive statistics are calculated including numbers, percentage, mean and standard deviation. Inferential statistics are analyzed with SPSS (version 22) to determine correlation between results of performance observation, Visual inspection and ATP interpretation by using Chi-square test or Fisher's exact test. The phi coefficient are calculated to measure strength between two sets of data. The phi coefficient refers to the meaning of Pearson's Correlation coefficients, values 0.01-0.19 as no or negligible, 0.2-0.39 as weak positive, 0.4-0.69 as medium positive, 0.7-1.0 as strong positive.12 The ATP readings were compared between "not compliant" and "compliant", and between "not clean" and "clean" respectively by using Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

rooms after patients are discharged

Exclusion Criteria:

no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rooms after patients are discharged
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of clean | immediately after terminal cleaning
  Free of dust, debris, and stains
rate of compliant | up to 10 hours (during cleaning practice)
  Surfaces were cleaned and disinfected properly
rate of pass | ten minutes after disinfection
  ATP readings less than 10 RLU

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chun Chen, MS, Principal Investigator — Taichung Veterans General Hospital Infection Control Center
Locations (1):
- Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No